CLINICAL TRIAL: NCT00674128
Title: Prospective Comparison of Cyanoacrylate Tissue Adhesive (Dermabond) and Suture (Vicryl) for Closure of Cardiac Device Pockets
Brief Title: Comparison of Cyanoacrylate Tissue Adhesive and Suture for Closure of Cardiac Device Pockets
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Mayo Clinic (Other)
Responsible Party: Gregory Altemose, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-001566
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Cardiovascular Disease
Keywords: pacemaker; cardioverter-defibrillator; ICD; cardiac resynchronization device; cyanoacrylate; suture; Dermabond; Vicryl
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhesive (Experimental): Cyanoacrylate tissue adhesive.
  Interventions: Device: Cyanoacrylate tissue adhesive (Dermabond)
- Suture (Active Comparator): Polyglactin 910 suture.
  Interventions: Device: Polyglactin 910 suture (Vicryl)

INTERVENTIONS:
Device: Cyanoacrylate tissue adhesive (Dermabond) — Skin closure will be performed with cyanoacrylate tissue adhesive.
  Other Names: Dermabond
  Arms: Adhesive
Device: Polyglactin 910 suture (Vicryl) — Skin closure will be performed with polyglactin 910 suture.
  Other Names: Vicryl
  Arms: Suture

SUMMARY:
The purpose of this study is to determine whether cyanoacrylate tissue adhesive is as effective as polyglactin 910 suture for surgical closure of cardiac device pockets.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for implantation of a pacemaker or ICD in the deltopectoral region at Mayo Clinic Hospital in Phoenix.

Exclusion Criteria:

* Allergy to one of the closure materials.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Altemose, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited sequentially at a tertiary care medical center between 2 June 2008 and 19 February 2009.
Pre-assignment Details: 33 patients did not meet inclusion criteria. 16 eligible patients did not consent. 103 patients were eligible and consented. 55 were assigned to Adhesive and 48 to Suture. The procedure was aborted for 5 patients in the Adhesive group and 4 patients in the Suture group.
Period: Overall Study
Arm/Group | Adhesive | Suture
Started | 50 | 44
Completed | 25 | 21
Not Completed | 25 | 23
Not completed — Withdrawal by Subject | 25 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adhesive | Suture | Total
Number analyzed (Participants) | 50 | 44 | 94
Age Continuous [Mean (Standard Deviation); unit: years] | 77 (10) | 77.6 (9.2) | 77 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Reported Here Are the Number of Participants With Devices That Developed Infection
Time Frame: Within 3 months after surgery.
Measure: Number; unit: participants
Arm/Group | Adhesive | Suture
Number analyzed (Participants) | 25 | 21
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 3 months
Description: No adverse event data were collected other than infection.
Arm/Group | Adhesive | Suture
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/25 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adhesive (N=25) | Suture (N=21)
Device Pocket Infection (Infections and infestations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes